CLINICAL TRIAL: NCT01307137
Title: Peer-lead and Telemedicine Activated Care (PACT) in Diabetes Prevention and Management
Brief Title: Peer-led and Telehealth Comparative Effectiveness Research (CER) Adoption for Diabetes Prevention and Management
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Florida Veterans Affairs Foundation for Research and Education (U.S. Federal Agency)
Responsible Party: Hermes Florez, MD, MPH, PhD, Miami VAMC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00915
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2011-01

CONDITIONS: Diabetes; Pre-diabetes
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance

ARMS (2):
- Telehealth (TAP) (Experimental)
  Interventions: Behavioral: Telehealth Intervention
- Peer-led care (PC) (Experimental)
  Interventions: Behavioral: Peer-led intervention

INTERVENTIONS:
Behavioral: Peer-led intervention — An expert patient in the peer-led intervention will provide effective support for patients and families to accelerate adoption of CER for diabetes prevention and management in the elderly. This will lead to better self-efficacy and clinical outcomes.
  Those veterans enrolled in the MOVE! and HARC programs that have showed success in management of weight and Diabetes will be offered to become peer-leaders.
  * Weight management success is defined as a loss of at least 5% of the weight since enrollment
  * Diabetes management will be defined as adequate control of HbA1c and/ or blood pressure and lipids.
  The potentials peer-leaders will have a pre-assessment test to evaluate diabetes prevention and management knowledge and motivation and support skills.
  Other Names: PC
  Arms: Peer-led care (PC)
Behavioral: Telehealth Intervention — Participants in the TAP group will receive mobile phones that will be programmed to monitor specific clinical parameters and promote adoption of CER on prevention and management of diabetes, with protocols developed in part based on the input from the focus groups. These devices display messages, tips, reminders and questions regarding healthy lifestyle and clinical parameters of diabetes, which will be developed using best practice guidelines. Participants will be asked to respond to the questions daily if they can. Also they are asked to provide their daily weight, blood pressure, and glucose levels (the later only for patients with diabetes).
  Other Names: TAP
  Arms: Telehealth (TAP)

SUMMARY:
The prevalence of obesity and diabetes in older adults is increasing. Because older adults are often portrayed as less likely to change long-standing health behaviors, health promotion in this age group has lagged behind others. In fact, little attention has been given to the importance of diabetes prevention in community-dwelling older adults through the implementation of programs that promote healthy nutrition, increase physical activity and improve self-management. The Diabetes Prevention Program (DPP), which demonstrated the benefit of modest weight loss on the reduction of diabetes risk (58% overall reduction with a 71% reduction in the older population), has yet to be translated into widespread public health practice.

The overall objective of this protocol is to implement evidence-informed, innovative interventions to increase adoption of findings from comparative effectiveness research (CER) for diabetes management and prevention in South Florida older veterans. Specifically, the proposed study will test the hypothesis that Peer-led Care alone (PC), or activated by technology (TechnAlert-Peer or TAP), is superior to traditional methods of information dissemination (Usual Care or UC) for adoption of CER on prevention and management of diabetes, leading to better self-efficacy and clinical outcomes.

The investigators will conduct a 12-month randomized controlled trial in older veterans with prediabetes and diabetes participating in one of the Healthy Aging Regional Collaborative programs. Primary outcomes include changes in self-efficacy, weight, and hemoglobin A1c. Secondary outcomes include changes in blood pressure, lipids, physical function, quality of life, and health care utilization and the evaluation of potential racial/ethnic disparities in the process of adoption of CER for prevention and management of diabetes.

This study is expected to accelerate the implementation of CER evidence for diabetes prevention, addressing health and economic challenges in the care of overweight and obese veterans.

DETAILED DESCRIPTION:
The prevalence of obesity and diabetes in older adults has increased during the past 20 years and will increasingly affect medical and social services, as well as costs over time. Because older adults are often portrayed as less likely to change long-standing health behaviors, health promotion in this age group has lagged behind others. In fact, little attention has been given to the importance of diabetes prevention and management in community-dwelling older adults.

A recent report of obesity diagnosis and care practice in the Veterans Health Administration showed that elderly patients were less likely to receive obesity-related education or counseling [Noel 2010]. Intentional weight loss in obese older adults has not been widely advocated by health care providers due to the perceived uncertainty of whether the benefits outweigh the risks. There is also a need to overcome the barriers to provide appropriate interventions on blood pressure, glucose, and lipid management tailored to the functionality of older adults.

The Diabetes Prevention Program (DPP) demonstrated the benefit of modest weight loss, through diet and exercise, on the reduction of diabetes risk in participants from all race/ethnic groups (58% overall reduction with a 71% reduction in the older population), leading to a delay of 4 years over a 10-year period in the onset of diabetes among those that received lifestyle intervention [DPP 2002, DPP 2009]. The DPP is considered a landmark study in comparative effectiveness research (CER), but it has yet to be translated into widespread public health practice.

South Florida provides a unique setting to accelerate the adoption of this CER evidence into practice and address the obesity and diabetes challenges of the aging population. There are more than 800,000 multi-ethnic residents age 60 and over, many of whom have one or more chronic diseases [CDC 2008]. A large number of older veterans with or at high-risk of diabetes currently receive care in the Miami VA Healthcare System.

Compelling scientific evidence exists that lifestyle change delays the onset of type 2 diabetes in high-risk persons. Lifestyle intervention can also lead to a reduction in cardiovascular risk factors in individuals with type 2 diabetes [Look AHEAD research group 2007]. However, few older adults succeed in achieving intentional weight loss through healthy diet and increased physical activity. Furthermore, some have argued that the current US health system is not prepared to deliver lifestyle interventions [Narayan 2004].

Several issues related to integration of lifestyle intervention in clinical practice have been raised. Currently, it is unknown whether other practicing professionals could deliver interventions in the community with efficacy similar to that of the interventionists of the DPP, who were trained in counseling on nutrition, exercise, and behavior modification. The investigators propose the use of telemedicine with applications in an interactive web-based system. This will allow participants to get just-in-time feedback from peers using targeted information on specific areas that need reinforcement to adopt healthy lifestyle and better self-management skills by older veterans. This will bolster the peer-participant interaction and make them more focused around areas where there are adoption gaps. This technology functions as a platform for social interaction that will lead to increase self-efficacy and better health outcomes.

The VA National Center for Health Promotion and Disease Prevention (NCP) developed the MOVE! weight management program based on the 1998/2000 Identification and Treatment of Overweight and Obesity in Adults Evidence Report. A major goal for the MOVE! program has been to reduce the prevalence of diabetes in veterans. Our long-term goal is to reduce the burden of obesity-related chronic diseases and promote healthy aging in older veterans through the implementation of best practices for prevention. The main objective of this project is to implement evidence-informed, innovative interventions to increase adoption of findings from comparative effectiveness research (CER) for diabetes management prevention in South Florida older veterans.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years and older
2. Enrolled in HARC program
3. Body mass index (BMI) ≥ 25 kg/m²
4. Diagnosed diabetes or prediabetes [ADA 2003 criteria] HbA1c ≥ 5.7%
5. Able to operate a telemedicine device, respond to text queries, and use his/her glucose meter, a blood pressure monitor, and a scale for daily weights

Exclusion Criteria:

1. End-stage illness
2. Anticipated survival less than 12 months
3. Imminent nursing home placement
4. Diagnosis of psychosis or significant cognitive impairment/dementia

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Compare changes in self-efficacy between participants receiving peer-led care (with or without TAP intervention) and those receiving UC over 12 months. | 12 months
Compare changes in weight and hemoglobin A1c between participants receiving peer-led care (with or without TAP intervention) and those receiving UC over 12 months. | 12 months

SECONDARY OUTCOMES:
Compare changes in weight, hemoglobin A1c, and self-efficacy between white-non-hispanics and minorities over 12 months. | 12 months
  Measure changes in blood pressure, lipids, physical function, quality of life, health care utilization (physician visits, emergency visits, and days in hospital) among racial minorities compared to non-minorities.
Compare changes in blood pressure, lipids, physical function, and quality of life among treatment groups (UC, PC, and TAP). | 12 months
Compare changes in health care utilization (physician visits, emergency visits, and days in hospital) among treatment groups (UC, PC, and TAP). | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Lisset Oropesa, MD, Study Director — Miami VAMC; Hermes J Florez, MD, Principal Investigator — Miami VAMC
Locations (2):
- United States (2):
  - Miami VAMC, Miami, Florida
  - University of Miami, Miami, Florida